CLINICAL TRIAL: NCT01565603
Title: Intolerance Mechanisms and Exercise Performance Limitation During a High Altitude Stay: Investigation of Sleep and Cerebral Responses
Brief Title: Sleep and Cerebral Responses to High Altitude
Acronym: VALLOT 2011
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Principal Investigator, AdministrateurDRC, Principal investigator, University Hospital, Grenoble
Other Study IDs: RCB 2011-A00071-40
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Acute Mountain Sickness; High Altitude Pulmonary Edema; High Altitude Cerebral Edema
Keywords: Hypoxia; Exercise; Sleep; Brain; Neuromuscular function; Heart
MeSH Terms: conditions — Altitude Sickness; Hypoxia; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Venous blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Mechanisms underlying high-altitude intolerance as well as exercise performance limitation in hypoxia still remain to be fully understood. Recent data suggest that sleep disturbances on one hand and cerebral perturbations on teh other hand may be key mechanisms. The investigators evaluated 12 healthy subjects at sea level and at 4400 m of altitude for 7 days in order to better describe sleep and cerebral responses. The investigators hypothesized that sleep and cerebral disturbances play a critical role for the developement of acute mountain sickness and for exercise performance limitation during acute high-altitude exposure.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 50 yrs old
* Male

Exclusion Criteria:

* Respiratory, cardiac, metabolic or neuromuscular diseases
* History of severe acute mountain sickness

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy young subjects
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2011-07; Primary Completion 2011-10 (Actual); Study Completion 2012-10 (Estimated)